CLINICAL TRIAL: NCT02153814
Title: Pilot Study on the Effect of Endometrial Injury in Patients Undergoing in Vitro Fertilization (IVF)
Brief Title: Endometrial Injury and in Vitro Fertilization Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Northwestern Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NW-STU00075489
Record Dates: First submitted 2013-12-17; First posted 2014-06-03 (Estimated); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Infertility
Keywords: Infertility; In vitro fertilization; Endometrial injury
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Sham Comparator): Will undergo sham procedure twice
  Interventions: Procedure: Sham procedure
- One Endometrial Scratch Procedure (Experimental): Will undergo one sham procedure and one endometrial scratch procedure
  Interventions: Procedure: Endometrial Scratch
- Two Endometrial Scratch Procedures (Experimental): Will undergo endometrial scratch procedure twice
  Interventions: Procedure: Endometrial Scratch

INTERVENTIONS:
Procedure: Endometrial Scratch — After cleansing the cervix with Betadine, the procedure will be performed using a 3mm endometrial sampling curette, with three passes made of the endometrium along the length of the fundus. Patients will be given the option to take ibuprofen 600mg one hour prior to the scheduled procedure. The first endometrial scratch procedure or sham procedure will be performed up to two weeks prior to expected menses, and the second endometrial scratch or sham procedure will be performed cycle day 5-11 of the stimulation cycle.
  Other Names: Endometrial biopsy; Endometrial injury; Endometrial pipelle
  Arms: One Endometrial Scratch Procedure; Two Endometrial Scratch Procedures
Procedure: Sham procedure — For the sham procedure, after cleansing the cervix with betadine, the endometrial sampling curette will be placed 2-3cm into the cervix without entering the uterine cavity
  Arms: Control

SUMMARY:
Infertility affects 1 in 7 couples worldwide. The most successful treatment is in vitro fertilization (IVF), a procedure where a woman's eggs are collected and fertilized with sperm to make embryos, which are then placed in the woman's uterus using a small catheter, a procedure called "embryo transfer." Unfortunately, pregnancy rates from IVF are less than 50%. Recently, several studies have shown dramatically improved pregnancy rates by grazing the innermost lining of the uterus (the endometrium) with a small flexible catheter weeks prior to embryo transfer. These studies were all performed outside the United States (U.S.) in women with multiple failed IVF attempts and did not investigate the mechanisms by which endometrial injury works. This study will be the first to evaluate the effect of endometrial injury on IVF success in all women undergoing IVF, including first IVF cycles, frozen embryo transfers, and donor eggs.

DETAILED DESCRIPTION:
Nationally, the percentage of in vitro fertilization (IVF) cycles resulting in pregnancy is still less than 50%, even in optimal patients. While failed implantation may be due to embryo factors, in recent years much attention has been given to the role of endometrial receptivity at the time of embryo transfer. There is abundant evidence in the literature showing that, in women with repeated implantation failures despite having high quality embryos, endometrial injury performed either in the follicular phase of the IVF cycle or late in the cycle preceding the treatment cycle increases IVF success rates, often more than doubling the pregnancy rate.

The mechanism of improved pregnancy rates after endometrial injury is currently unknown. There is a paucity of studies in the current literature linking the biochemical and genetic changes induced by endometrial injury to pregnancy rates in patients undergoing IVF, as well as studies examining the effect of endometrial injury on ultrasound findings previously shown to predict IVF success, such as endometrial thickness, pattern, and volume, or markers of endometrial vascularity.

Additionally, no studies have been published examining whether or not IVF success rates can be improved in all-comers (not just women with repeated failures or abnormal appearing endometrium on ultrasound) by performing endometrial injury and there are currently no studies published on this topic with U.S. women in the study population. The proposed study would be the first to examine the effect of endometrial injury in U.S. women undergoing infertility treatment with IVF, regardless of prior treatment history, including women undergoing donor oocyte IVF cycles or frozen embryo transfer. It would also be the first to evaluate the biochemical changes induced by endometrial injury in the context of cycle outcome and live birth rate and to examine the effect on ultrasound parameters.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing IVF at the Northwestern Medical Faculty Foundation, Division of Reproductive Endocrinology and Infertility
* Age at time of egg retrieval 18-40 years, inclusive. Age at time of embryo transfer 18-45 years, inclusive.
* All subjects must have given signed, informed consent prior to registration in study

Exclusion Criteria:

* Patients with any current uterine pathology known to affect implantation, such as large hydrosalpinx, Asherman's syndrome, fibroids or polyps
* Patients with active cervical or pelvic infection
* Pregnant women
* Patients with a serious bleeding diathesis (e.g. hemophilia)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Actual)
Dates: Start 2014-08; Primary Completion 2017-06 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Live Birth Rate | 10 Months

SECONDARY OUTCOMES:
Pregnancy Rate | 2 months
Implantation Rate | 1 month
Spontaneous Abortion Rate | 4 months
3-D Ultrasound Results - endometrial volume in mm^3 | 1 month
Endometrial tissue gene expression levels (CT values) | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Erica E Marsh, MD, MSCI, Principal Investigator — Northwestern University; Molly B Moravek, MD, MPH, Study Director — Northwestern University; Randall Barnes, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Medical Faculty Foundation, Division of Reproductive Endocrinology and Infertility, Chicago, Illinois, United States